CLINICAL TRIAL: NCT00232219
Title: Use of Fish Oils to Reduce Recurrence of Atrial Fibrillation Following DC Cardioversion.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003.188
Record Dates: First submitted 2005-10-02; First posted 2005-10-04 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fish Oils

ARMS (2):
- Control (No Intervention): No fish oil exposure
- Fish oil (Experimental): Patients given 6g/day of fish oil containing 1.8g/d of EPA+DHA in a 1.5:1 ratio.
  Interventions: Drug: Fish oil

INTERVENTIONS:
Drug: Fish oil
  Arms: Fish oil

SUMMARY:
The purpose of this study is to investigate whether fish oil supplements may be beneficial in preventing the recurrence of atrial fibrillation after cardioversion.

Atrial fibrillation is a heart condition which can sometimes be successfully treated by a cardioversion.

Cardioversion involves resetting the heart back to normal with the use of electric current.

There is a tendency for the atrial fibrillation to recur , days weeks or even months after the cardioversion.

Fish oil supplements may be of benefit to patients with heart problems Recent evidence suggests that fish oils may be beneficial to patients with rhythm disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent Atrial Fibrillation on Warfarin.

Exclusion Criteria:

* paroxysmal atrial fibrillation with self terminating episodes.
* left atrial size>6.0cm
* myocardial infarction in the previous 6 months.
* contraindications to amiodarone use .
* cardiac surgery in the previous 3 months .
* an acute reversible illness contributing to the development of af
* a QTc interval > 480ms.
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation followed cardioversion | 1 year

OTHER OUTCOMES:
Safety and tolerability | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sparks, MBBS, PhD. FRACP, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne hospital, Melbourne, Victoria, Australia